CLINICAL TRIAL: NCT05736185
Title: Effect of Electric Impedance Tomography-Guided PEEP Titration on the Ventilation-perfusion Mismatch in Moderate or Severe ARDS
Brief Title: Effect of Electric Impedance Tomography-Guided PEEP Titration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EIT-PEEPstudy
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EIT-PEEP strategy (Experimental): PEEP selected by EIT which remained at 15 min
  Interventions: Device: PEEP selection
- Low FiO2-PEEP strategy (Experimental): PEEP selected by low FiO2-PEEP table which remained at 15 min
  Interventions: Device: PEEP selection
- High FiO2-PEEP strategy (Experimental): PEEP selected by high FiO2-PEEP table which remained at 15 min
  Interventions: Device: PEEP selection

INTERVENTIONS:
Device: PEEP selection — Electric impedance tomography-guided PEEP titration

SUMMARY:
Acute respiratory syndrome distress (ARDS) is a clinical common syndrome with high mortality. Mechanical ventilation (MV) is the cornerstone of management of ARDS but can lead to ventilator-induced lung injury. Positive end-expiratory pressure (PEEP), as one of main component of MV, has been widely used in the clinical practice. However, how to best set PEEP is still a difficult problem for moderate to severe ARDS patients. EIT, an imaging tool evaluating the regional ventilation distribution at the bedside, can achieve the individual PEEP selection for all mechanically ventilated patients. This article compared the effect of PEEP titrated guided by EIT with fraction of inspired oxygen (FiO2)-PEEP table on the ventilation-perfusion mismatch.

ELIGIBILITY:
Inclusion Criteria:

1. Intubated patients with moderate and severe ARDS (Berlin definition, PaO2/FiO2 ≤200 mmHg at PEEP 5 cmH2O)
2. undergoing deep sedation on controlled mechanical ventilation within72 hours after ARDS onset

Exclusion Criteria:

1. age <18 years old
2. patient undergoing legal protection
3. contra-indications to EIT (e. g. severe chest trauma or wounds)
4. pneumothorax
5. patient undergoing ECMO
6. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Difference in ventilation-perfusion mismatch between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  EIT-PEEP was obtained by EIT, low-PEEP was obtained by low FIO2-PEEP table, and high-PEEP was obtained by high FIO2-PEEP table.

SECONDARY OUTCOMES:
difference in center of ventilation (COV) between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  COV was obtained by EIT monitoring
Difference in dead space measured with EIT between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  dead space was obtained by EIT monitoring
Difference in shunt measured with EIT between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  shunt was obtained by EIT monitoring
Difference in wasted ventilation measured with EIT between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  wasted ventilation was obtained by EIT monitoring
Difference in wasted perfusion measured with EIT between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  wasted perfusion was obtained by EIT monitoring
ventilation distribution measured with EIT between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  ventilation distribution was obtained by EIT in difference regions
perfusion distribution measured with EIT between EIT-PEEP, low-PEEP, and high PEEP | up to 24 hours
  perfusion distribution was obtained by EIT in difference regions
Correlations between ventilation-perfusion mismatch and overdistension and lung collapses | up to 24 hours
  Overdistension (%) and lung collapses (%) will be assessed by EIT. These two values cannot be measured separately. V/Q mismatch will be computed by EIT, and expressed in %. Correlation will be performed by linear regression.
recruitment-to-inflation (R/I) ratio | up to 24 hours
  recruitment-to-inflation (R/I) ratio was computed between the two PEEP levels
PaO2/FIO2 | up to 24 hours
  PaO2/FIO2 was obtained by gas analysis
respiratory system mechanics | up to 24 hours
  respiratory system compliance included lung compliance, chest wall compliance, and respiratory system compliance. respiratory system resistance will be computed as the inverse of compliance.
Correlation between V/Q mismatch markers and recruitability | up to 24 hours
  Recruitability will be assessed between 15 and 5 cmH2O by respiratory mechanics, as the recruited volumes value (in mL). R/I ratio will be derived from these data (no unit). V/Q mismatch will be computed by EIT, and expressed in %. Correlation will be performed by linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: liu ling, phD, Study Director — Zhongda Hospital, School of Medicine, Southeast University
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No